CLINICAL TRIAL: NCT00843583
Title: A Cross-sectional Study of the Occurrence and Effect of Obstructive Sleep Apnea in Subjects With Resistant Hypertension
Status: Completed | Type: Observational
Sponsor: The University of Hong Kong (Other)
Responsible Party: Professor Ip, Sau Man Mary, Department of Medicine, The University of Hong Kong, Queen Mary Hospital
Other Study IDs: NCT00843583
Record Dates: First submitted 2009-02-12; First posted 2009-02-13 (Estimated); Last update posted 2017-05-03 (Actual); Status verified 2017-05

CONDITIONS: Obstructive Sleep Apnea; Resistant Hypertension
Keywords: prevalence; obstructive sleep apnea; resistant hypertension
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Blood test for glucose, lipid, vascular and metabolic markers
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- resistant hypertension subjects: subjects with resistant hypertension

SUMMARY:
This study aims to investigate the prevalence of obstructive sleep apnea (OSA) in subjects with resistant hypertension and to evaluate the relationship between parameters of OSA severity and blood pressure control

DETAILED DESCRIPTION:
Obstructive sleep apnea (OSA) is characterized by intermittent upper airway collapse during sleep, which results in hypoxia, arousals and surge in sympathetic activity. There is robust evidence to support a contributing role of OSA in hypertension (HT). The Sleep Heart Health Study (1), which recruited more than 6000 subjects having polysomnogram at home, found an independent association between OSA and HT. The adjusted odds ratio was 1.37 for subjects with and apnea-hypopnea index >= 30/hour compared to those without apnea. The Wisconsin Sleep Cohort Study , which provided prospective longitudinal follow-up for OSA subjects over 4 years, have shown dose dependency of the severity of OSA and the risk of development of HT. Current available data suggests that in hypertensive patients with severe OSA, there is a BP drop of about 10mmHg with CPAP treatment (2-5). The blood pressure (BP) lowering effect of CPAP treatment in the group with mild asymptomatic OSA is less consolidated.

The relationship between BP and risk of cardiovascular events is continuous, consistent, and independent of other risk factors. A strict blood pressure control is imperative in subjects with diabetes mellitus or renal impairment. Resistant hypertension is defined as blood pressure that remains above goal in spite of concurrent use of 3 antihypertensive agents of different classes. (6) Resistant hypertension is defined in order to identify patients who are at risk of having secondary causes of hypertension, and who may benefit from specific diagnostic and therapeutic applications. Despite the fact that OSA is listed as one of the causes of resistant HT (6), paucity of works has demonstrated the scale of problems of untreated OSA in subjects with resistant HT. (7-9) There is so far one study demonstrating the beneficial effect of CPAP treatment in subjects with resistant HT, though no randomization was implemented and the sample size was limited (n=11). (10) We aim at conducting a cross-sectional study to explore the situation which would guide further clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* ≧ 3 anti-HT drugs
* age 18-65
* mentally fit for signing an informed written consent

Exclusion Criteria:

* moderate renal impairment (glomerular filtration rate <30 mL/min/m2 )
* endocrine/renal/cardiac causes of secondary HT
* congestive heart failure and clinically fluid overloaded
* On drugs that elevate BP e.g. alcohol, NSAID, steroid

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive sampling of subjects who attend Hypertension clinic , Department of Medicine, Queen Mary Hospital, and who fulfill the inclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 96 (Estimated)
Dates: Start 2009-02; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
ambulatory blood pressure | 24 hour

CONTACTS AND LOCATIONS:
Overall Officials: Sau Man Mary Ip, MD, Principal Investigator — Department of Medicine, The University of Hong Kong
Locations (1):
- Department of Medicine, The University of Hong Kong, Queen Mary Hospital, Hong Kong, Hong Kong

REFERENCES:
- [Background] Nieto FJ, Young TB, Lind BK, Shahar E, Samet JM, Redline S, D'Agostino RB, Newman AB, Lebowitz MD, Pickering TG. Association of sleep-disordered breathing, sleep apnea, and hypertension in a large community-based study. Sleep Heart Health Study. JAMA. 2000 Apr 12;283(14):1829-36. doi: 10.1001/jama.283.14.1829. PMID 10770144
- [Background] Pepperell JC, Ramdassingh-Dow S, Crosthwaite N, Mullins R, Jenkinson C, Stradling JR, Davies RJ. Ambulatory blood pressure after therapeutic and subtherapeutic nasal continuous positive airway pressure for obstructive sleep apnoea: a randomised parallel trial. Lancet. 2002 Jan 19;359(9302):204-10. doi: 10.1016/S0140-6736(02)07445-7. PMID 11812555
- [Background] Becker HF, Jerrentrup A, Ploch T, Grote L, Penzel T, Sullivan CE, Peter JH. Effect of nasal continuous positive airway pressure treatment on blood pressure in patients with obstructive sleep apnea. Circulation. 2003 Jan 7;107(1):68-73. doi: 10.1161/01.cir.0000042706.47107.7a. PMID 12515745
- [Background] Mills PJ, Kennedy BP, Loredo JS, Dimsdale JE, Ziegler MG. Effects of nasal continuous positive airway pressure and oxygen supplementation on norepinephrine kinetics and cardiovascular responses in obstructive sleep apnea. J Appl Physiol (1985). 2006 Jan;100(1):343-8. doi: 10.1152/japplphysiol.00494.2005. PMID 16357087
- [Background] Norman D, Loredo JS, Nelesen RA, Ancoli-Israel S, Mills PJ, Ziegler MG, Dimsdale JE. Effects of continuous positive airway pressure versus supplemental oxygen on 24-hour ambulatory blood pressure. Hypertension. 2006 May;47(5):840-5. doi: 10.1161/01.HYP.0000217128.41284.78. Epub 2006 Apr 3. PMID 16585412
- [Background] Calhoun DA, Jones D, Textor S, Goff DC, Murphy TP, Toto RD, White A, Cushman WC, White W, Sica D, Ferdinand K, Giles TD, Falkner B, Carey RM. Resistant hypertension: diagnosis, evaluation, and treatment. A scientific statement from the American Heart Association Professional Education Committee of the Council for High Blood Pressure Research. Hypertension. 2008 Jun;51(6):1403-19. doi: 10.1161/HYPERTENSIONAHA.108.189141. Epub 2008 Apr 7. PMID 18391085
- [Background] Logan AG, Perlikowski SM, Mente A, Tisler A, Tkacova R, Niroumand M, Leung RS, Bradley TD. High prevalence of unrecognized sleep apnoea in drug-resistant hypertension. J Hypertens. 2001 Dec;19(12):2271-7. doi: 10.1097/00004872-200112000-00022. PMID 11725173
- [Background] Grote L, Hedner J, Peter JH. Sleep-related breathing disorder is an independent risk factor for uncontrolled hypertension. J Hypertens. 2000 Jun;18(6):679-85. doi: 10.1097/00004872-200018060-00004. PMID 10872551
- [Background] Lavie P, Hoffstein V. Sleep apnea syndrome: a possible contributing factor to resistant. Sleep. 2001 Sep 15;24(6):721-5. doi: 10.1093/sleep/24.6.721. PMID 11560187
- [Background] Logan AG, Tkacova R, Perlikowski SM, Leung RS, Tisler A, Floras JS, Bradley TD. Refractory hypertension and sleep apnoea: effect of CPAP on blood pressure and baroreflex. Eur Respir J. 2003 Feb;21(2):241-7. doi: 10.1183/09031936.03.00035402. PMID 12608436
- [Derived] Lui MMS, Tse HF, Mak JCW, Lam DCL, Chan CWS, Chong PWC, Ip MSM. Untreated Obstructive Sleep Apnea Is Associated With Myocardial Injury Independent of Blood Pressure Control in Hypertension. J Clin Sleep Med. 2018 Nov 15;14(11):1841-1847. doi: 10.5664/jcsm.7476. PMID 30373683